CLINICAL TRIAL: NCT05151146
Title: A Phase 1 Study to Investigate the Pharmacokinetics of ANJ900 (Metformin Hydrochloride Delayed-release Tablets) and the Effect of Food on the Pharmacokinetics of ANJ900 in Chinese Healthy Subjects
Brief Title: A Phase 1 Study of ANJ900 Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anji Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANJ900D1104
Record Dates: First submitted 2021-11-16; First posted 2021-12-09 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ANJ900 in the fasted state (Experimental): Single dose (1800 mg) of ANJ900
  Interventions: Drug: ANJ900
- ANJ900 in the fed state (Experimental): Single dose (1800 mg) of ANJ900
  Interventions: Drug: ANJ900
- Metformin IR in the fasted state (Active Comparator): Single dose (1000 mg) of metformin IR
  Interventions: Drug: Metformin IR

INTERVENTIONS:
Drug: ANJ900 — Metformin hydrochloride delayed-release tablets
  Other Names: Met DR
  Arms: ANJ900 in the fasted state; ANJ900 in the fed state
Drug: Metformin IR — metformin hydrochloride
  Other Names: Met IR
  Arms: Metformin IR in the fasted state

SUMMARY:
This will be a Phase 1, randomised, open label, 3 way crossover study in healthy male and female Chinese subjects. Subjects will participate in 3 treatment periods and will be randomised in a 1:1:1 ratio to 1 of 3 treatment sequences. There will be a washout period of 7 days between doses.

DETAILED DESCRIPTION:
This will be a Phase 1, randomised, open label, 3 way crossover study in healthy male and female Chinese subjects. Subjects will participate in 3 treatment periods and will be randomised in a 1:1:1 ratio to 1 of 3 treatment sequences. There will be a washout period of 7 days between doses.

All subjects will receive each of the following treatments:

* Treatment 1: A single dose of 1800 mg ANJ900 in the fasted state.
* Treatment 2: A single dose of 1800 mg ANJ900 in the fed state.
* Treatment 3: A single dose of 1000 mg metformin IR in the fasted state. Potential subjects will be screened to assess their eligibility to enter the study within 14 days prior to the first dose administration. Subjects will be admitted into the study site on Days 1, 7, and 14 and will be confined to the study site until discharge on Days 3, 10, and 17 respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese males or females between 18 and 65 years of age, inclusive.
2. Body mass index between 18.5 and 28.0 kg/m2, inclusive, with a body weight >50 kg (males) or >45 kg (females).
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG (including heart rate ≥50 bpm, PR interval <200 ms, and QRS duration <120 ms), vital signs measurements (systolic blood pressure ≥90 and <140 mmHg and diastolic blood pressure ≥50 and <90 mmHg), and clinical laboratory evaluations at screening and Day -1 as assessed by the investigator (or designee).
4. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception as detailed in Appendix 3.
5. Able to comprehend and willing to sign an ICF, remain at the study site, and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic (eg, asthma, urticaria, eczema dermatitis), dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
2. Malignancy within 5 years (except basal cell skin carcinoma).
3. History of a clinically significant disease that affects drug absorption, metabolism, or elimination processes, as determined by the investigator (or designee), including, but not limited to:

   1. inflammatory bowel disease, gastritis, ulcers, bile duct stones, or internal bleeding of the gastrointestinal tract or rectum
   2. gastrointestinal surgery (eg, anastomosis or bowel resection)
   3. pancreatic injury or pancreatitis
   4. urinary tract obstruction or difficulty passing urine.
4. History of hypoglycaemic episodes, severe unconscious hypoglycaemia, or glucose metabolism disorders.
5. History of significant hypersensitivity, intolerance, or allergy to any drug compound (eg, metformin), food, or other substance, unless approved by the investigator (or designee).
6. Active symptoms, or a recent diagnosis of, coronavirus disease-19 (COVID-19).
7. Donation or loss of >500 mL of blood within 4 weeks prior to screening.
8. Receipt of blood products within 8 weeks prior to screening.
9. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months.
10. Poor peripheral venous access or intolerant of venous blood collection.
11. Use or intend to use any prescription medications (with the exception of paracetamol [≤4000 mg/day] or ibuprofen [≤2400 mg/day]) within 4 weeks or 5 half lives, whichever is longer, prior to screening.
12. Use or intend to use any over the counter medications (with the exception of paracetamol [≤4000 mg/day], ibuprofen [≤2400 mg/day], and topical over the counter medications for external use), herbal medications, or food supplements (eg, vitamins or mineral supplements) within 2 weeks or 5 half lives, whichever is longer, prior to screening.
13. Fasting plasma glucose <3.9 mmol/L or >6.1 mmol/L at screening or Day -1.
14. Alanine aminotransferase, aspartate aminotransferase, or direct bilirubin >1.5 × the upper limit of normal at screening or Day -1.
15. Positive hepatitis panel, human immunodeficiency virus test, or syphilis test.
16. History of alcoholism or drug/chemical abuse within 12 months.
17. Alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
18. Have consumed foods and beverages containing caffeine, xanthine, alcohol, or components that affect the absorption, metabolism, and excretion of drugs (eg, grapefruit or Seville oranges) within 48 hours prior to check-in.
19. Have smoked >5 cigarettes or use the equivalent tobacco or nicotine containing products per day in the past 3 months, or are unwilling to abstain from smoking cigarettes or use the equivalent tobacco or nicotine containing products from 48 hours prior to Day -1 until discharge.
20. Are unwilling to abstain from strenuous exercise from 48 hours prior to Day -1 until discharge.
21. Positive alcohol breath test, urine drugs of abuse test, or urine cotinine test.
22. Subjects who, in the opinion of the investigator (or designee), should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Characterize the AUC of single oral dose of ANJ900 in healthy Chinese subjects | 1 week
  ANJ900 levels in blood will be collected in serial draws
Characterize Cmax of a single oral dose of ANJ900 in healthy Chinese subjects | 1 week
  ANJ900 levels in blood will be collected in serial draws

SECONDARY OUTCOMES:
Characterize the urine excretion from time zero to 24 hours post does of metformin | 1 week
  Urine will be analyzed for ANJ900
Assess the safety of ANJ900 in healthy Chinese subjects | 3 weeks
  Adverse events will be collected and reported

CONTACTS AND LOCATIONS:
Overall Officials: Dongyang Liu, MD, Principal Investigator — Peking University Third Hospital; Haiyan Liu, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Haidan, China

IPD SHARING:
Plan to Share IPD: No